CLINICAL TRIAL: NCT06610903
Title: Study Protocol for a Single-center, Randomized, Open-label, Two-formulation, Single-dose, Two-cycle, Double-crossover Fasting Bioequivalence Trial of Hemay005 Tablets in Healthy Subjects
Brief Title: Bioequivalence Test of Hemay005 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HM005PS1S09
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Hemay005

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subject group 1 (Experimental): 15mg/tablet，one tablet each time. Participants will receive a single dose of Hemay005 tablet in Day1and Day8
  Interventions: Drug: Hemay005
- Healthy subject group 2 (Experimental): 15mg/tablet，one tablet each time. Participants will receive a single dose of Hemay005 tablet in Day1and Day8
  Interventions: Drug: Hemay005

INTERVENTIONS:
Drug: Hemay005 — In the first cycle, 15mg (1 tablet/person) was given on an empty stomach for Hemay005-T1 or Hemay005-T2, and the second cycle was crossed over

SUMMARY:
The pharmacokinetics behavior of the test formulation T1 and the control formulation T2 were evaluated by oral administration in healthy subjects under fasting state to evaluate the bioequivalence of the two formulations.

DETAILED DESCRIPTION:
To evaluate the pharmacokinetics and bioequivalence of the test formulation T1 and the control formulation T2 in healthy subjects under fasting state. The safety of the two preparations in vivo was observed

ELIGIBILITY:
Inclusion Criteria:

* male and female subjects aged from 18 to 65 years old (including 18 and 65 years old), with an appropriate gender ratio;
* body weight: no less than 50.0kg for men, no less than 45.0kg for women, and body mass index (BMI) [= weight (kg)/height 2 (m2)] between 19.0 and 26.0 kg/m2 (including boundary values);
* 90mmHg≤ systolic blood pressure <140mmHg, 60mmHg≤ diastolic blood pressure <90 mmHg, 60 BPM ≤ pulse ≤100 BPM, normal body temperature;
* have understood the nature, significance, possible benefits, possible inconvenience and potential risks of the trial in detail before the trial, and voluntarily participate in the clinical trial, can communicate well with the investigators, comply with the requirements of the whole study, and sign the written informed consent.

Exclusion Criteria:

* Participants who participated in clinical trials of other drugs/devices within 3 months and used the investigational drugs/devices;
* (Inquiry) patients with abnormal clinical manifestations that need to be excluded, including but not limited to diseases of the nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal system, respiratory system, metabolic system, skeletal system and other systems;
* (inquiry) the history of vomiting, diarrhea or any physiological condition that could interfere with the test results within 7 days before the test;
* (Enquire) patients with specific allergic history (asthma, urticaria, eczema, etc.), or allergic to any drug, food or pollen, or known allergic to PDE4 inhibitors (e.g., apemilast, roflumilast, etc.);
* (inquiry) those who have lost blood or donated more than 400mL of blood within 3 months before the trial, or intend to donate blood during the trial;
* (Inquiry) pregnant or lactating women, or subjects (including male subjects) who have fertility or sperm or egg donation plans from 30 days before the study to 6 months after the last dose of the study, and who are unwilling or unable to use effective contraceptive measures;
* general physical examination and laboratory tests (blood routine, blood biochemistry, coagulation function, urine routine, stool routine, blood/urine pregnancy (female), etc.) within 7 days before the test, and electrocardiogram (ECG) results judged by clinicians as clinically significant within 14 days before the test;
* if one or more of hepatitis B virus surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody or treponema pallidum antibody is clinically significant;
* (inquiry) patients who had a clinically significant major disease or underwent a major surgical operation within 3 months before the trial;
* (inquiry) Subjects who consumed more than 14 units of alcohol per week (1 unit = 17.7 mL ethanol, i.e. 1 unit = 354 mL of 5% beer or 44mL of 40% liquor or 147 mL of 12% wine) in the 3 months before the trial, or who could not abstain from alcohol during the trial;
* (Inquired) smoked more than 5 cigarettes per day in the 3 months before the trial, or could not stop using any tobacco products during the trial;
* (inquiry) consuming excessive amounts of tea, coffee and/or caffeine-rich beverages (> 8 cups, 1 cup =250 mL) per day in the 3 months before the study;
* (question) consumed any foods or drinks (such as strong tea, coffee, chocolate, cola, animal organs, grapefruit, dragon fruit, mango, etc.) rich in caffeine/xanthine or other special ingredients (such as strong tea, coffee, chocolate, cola, animal organs, grapefruit, dragon fruit, mango, etc.) from screening to -2 days of admission, or could not stop eating the above foods or drinks during the study;
* (inquiry) use of any drugs that inhibit or induce hepatic drug-metabolizing enzymes (e.g., inducers - barbiturates, carbamazepine, phenytoin, glucocorticoids; Inhibitors (SSRI antidepressants, cimetidine, sedative- hypnotics, verapamil, fluoroquinolones, antihistamines);
* (inquiry) those who are unable to eat or have swallowing difficulties, have special dietary requirements and/or cannot follow a uniform diet;
* (inquirers) with a history of asthma or seizures;
* (inquired) who had used any prescription drugs, over-the-counter drugs, nutricals, herbal products or received vaccines within 14 days before the trial;
* (Inquiry) Mechanical operators who are engaged in high-altitude work, motor vehicle driving and other associated hazards;
* (inquiry) can not tolerate venipuncture and/or have a history of dizziness;
* (asked) who had used any drugs in the year before the test;
* alcohol breath test results > 0.0mg/100mL or drug abuse screening positive (morphine, methamphetamines, ketamine, dimethylenedioxyamphetamine, tetrahydrocannabinol acid, cocaine);
* subjects who were considered by the investigator to have poor adherence or any factor that precluded participation in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Relevant pharmacokinetic parameters，Peak Plasma Concentration（Cmax） | Day1-4，Day8-11
  All subjects who receive the drug will be analyzed for pharmacokinetic
Relevant pharmacokinetic parameters，Area under the plasma concentration versus time curve（AUC0-t） | Day1-4，Day8-11
  All subjects who receive the drug will be analyzed for pharmacokinetic
Relevant pharmacokinetic parameters，Area under the curve from time 0 extrapolated to infinite time (AUC0-inf) | Day1-4，Day8-11
  All subjects who receive the drug will be analyzed for pharmacokinetic

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Central Hospital, Wuhan, Hubei, China